CLINICAL TRIAL: NCT00060866
Title: Propranolol for Syncope With Sympathoadrenal Imbalance
Brief Title: Propranolol to Treat Fainting Due to Sympathoadrenal Imbalance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030182; 03-N-0182
Record Dates: First submitted 2003-05-14; First posted 2003-05-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Neurocardiogenic Syncope
Keywords: Beta-Adrenoceptors; Beta-Adrenoceptor Blocker; Neurocardiogenic Syncope; Chronic Orthostatic Intolerance; Neurocardiogenic; Dysautonomia; Autonomic Nervous System; Nurocardiogenic Syncope; NCS; Sympathoadrenal Imbalance; SAI; Orthostatic Intolerance
MeSH Terms: conditions — Syncope, Vasovagal; Autonomic Nervous System Diseases; Orthostatic Intolerance | interventions — Propranolol

INTERVENTIONS:
Drug: Propranolol

SUMMARY:
This study will examine the effectiveness of the drug propranolol in preventing fainting in patients with sympathoadrenal imbalance (SAI). SAI is a particular pattern of nervous system and chemical responses in which the blood vessels in skeletal muscles do not remain constricted appropriately during standing for a long time. This can lower blood pressure and cause fainting. Propranolol Inderal (registered trademark) is a Food and Drug Administration-approved drug that belongs to a class of drugs called beta-blockers. These drugs slow the heart rate and maintain blood pressure in certain situations.

Patients 18 years of age and older with SAI may be eligible for this study. Screening includes a tilt table test, described below, to determine if the patient has a particular chemical pattern in the blood.

Patients enrolled in the study take propranolol pills in increasing doses during the first week of the study to determine the proper dose for the individual. Then, the drug is stopped until the experimental phase of the study begins. In this phase, patients are randomly assigned to take either propranolol or placebo (look-alike pill with no active ingredient) for 4 days. On the fourth day, the patient undergoes a tilt table test to determine whether the treatment affects the patient's ability to tolerate tilt. For this test, the patient lies on a padded table with a motorized tilt mechanism that can move the patient from a flat position to an upright position in about 10 seconds. The patient remains upright for up to 45 minutes while the following measurements are taken:

* Arterial blood pressure monitoring and arterial blood sampling. A catheter (thin, plastic tube) is inserted into an artery in the elbow crease area of the arm or the wrist. This catheter allows continuous blood pressure monitoring and sampling of arterial (oxygenated) blood during the tilt test.
* Venous blood sampling and measurement of epinephrine and norepinephrine release. A catheter is inserted into a vein in each arm, one to collect venous (deoxygenated) blood samples, and the other to inject radioactive epinephrine (adrenaline) and norepinephrine (noradrenaline). These radioactive drugs, or ,tracers, allow measurement of the rate of release of the body's own norepinephrine and epinephrine into the bloodstream.
* Physiologic measurements. Blood pressure, heart rate, and EKG are measured continuously during the tilt test session, and blood flows and skin electrical conduction are measured intermittently. Blood flow is measured using sensors applied to the skin and a blood pressure cuff around the limb. For skin blood flow measurements, a laser beam scans the skin surface. The skin electrical conduction test measures how well the skin conducts electricity. This is measured through sensors placed on the fingers or other sites.

The effects of the test drug are allowed to wear off for 1 week, after which the entire tilt test procedure is repeated. Patients who were given propranolol for the first test session take placebo for the repeat session, and those who were given placebo take propranolol.

DETAILED DESCRIPTION:
This protocol is to evaluate treatment with oral propranolol for a particular form of neurocardiogenic syncope (NCS), characterized by a neuroendocrine pattern called, sympathoadrenal imbalance, (SAI). In SAI, plasma epinephrine levels increase progressively and to a greater extent than do plasma norepinephrine levels, before development of NCS. The SAI pattern is associated with skeletal muscle vasodilation, which also precedes NCS. We hypothesize that increased occupation of beta-2 adrenoceptors in skeletal muscle by high circulating epinephrine levels precipitates a neurocirculatory positive feedback loop leading to NCS. In this protocol we test this hypothesis using the non-selective beta-adrenoceptor blocker, propranolol. We predict that in patients with previously documented SAI and tilt-evoked NCS, propranolol treatment will improve orthostatic tolerance during follow-up tilt table testing, in a randomized, crossover-design, placebo-controlled, double-blind trial. The main department measures are occurrence of tilt-induced NCS, duration of tilt tolerance, hemodynamic and neurochemical indices of SAL, and patient questionnaire reports.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects are patients referred for evaluation of chronic orthostatic intolerance. Patients enter into the therapeutic trial after they are determined to have NCS with SAI in a screening evaluation. Participation in this protocol is offered to individuals 18 years old or older, independently of gender, race, advanced age, ethnicity, religion, or any demographic or sociopolitical classifications.

EXCLUSION CRITERIA:

Age: Minors younger than 18 years old are excluded. Advanced age does not constitute an exclusion criterion.

Risk: A candidate subject is excluded if, in the judgement of the Principal Investigator or Clinical Director, protocol participation would place the subject at subject at substantially increased acute medical risk. This includes the risks associated with air travel to the NIH. A candidate subject is excluded if, in the opinion of the Principal Investigator or Clinical Director, the medical risk outweighs the potential scientific benefit.

Disqualifying Conditions: A candidate subject is excluded if there is a disqualifying condition. Examples of disqualifying conditions are history of asthma or chronic obstructive pulmonary disease requiring bronchodilators, hepatic or renal failure, atrioventricular block of any degree, bradycardia, symptomatic congestive heart failure, severe anemia, psychosis, refractory ventricular arrhythmias, symptomatic coronary heart disease, insulin-dependent diabetes mellitus, Wolff-Parkinson-White syndrome, and peripheral vascular disease. Patients with known or suspected allergy or hypersensitivity to propranolol are excluded from this study. A positive HIV test result does not necessarily exclude a patient from participating.

Medications: A candidate subject is excluded if clinical considerations require that the patient continue treatment with a drug likely to interfere with the scientific results. Patients who must take medications daily in the following categories are excluded: anticoagulants, tricyclic, antidepressants, barbiturates, aspirin, acetaminophen, insulin, bronchodilators. Patients unable to discontinue nicotine, caffeine, or alcohol temporarily are excluded. Patients with chronic alcohol intake are excluded. Patients are not to discontinue any medications before the patient or the patient's doctor discusses this with the Principal Investigator, an Associate Investigator, or Research Nurse. If it is decided that discontinuing medications would be unsafe, then the patient is excluded from the study.

Herbal Medicines and Dietary Supplements: Certain herbal medicines or dietary supplements are known or suspected to interfere with the experimental results, and such herbal medicines or dietary supplements must be discontinued before enrollment in the study. For many herbal medicines or dietary supplements, the mechanisms of action and therefore the possible effects on the experimental results are unknown. In cases where the subjects wish to continue their herbal medicines or dietary supplements while on study, and search of the available medical literature fails to identify effects that are known or expected to interfere with the experimental results, then the subjects may participate.

Practical Limitations: Patients in whom we feel it would be difficult to technically to carry out the testing procedures are excluded.

Pregnancy: Pregnant or lactating women are excluded. A blood test for pregnancy will be conducted on women of childbearing potential, before intake evaluation and also before each drug treatment phase. During the course of the protocol, subjects who are women of childbearing potential will be advised to practice adequate contraception.

Termination of Participation: Subjects may refuse certain tests or procedures, or may terminate participation early, without loss of benefits to which they were previously entitled. The Investigators may also exclude a subject from further participation, such as in the event of known or suspect falsification of medical history information or refusal to undergo planned tests or procedures, without loss of benefits to which the subject was previously entitled.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 2003-05; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Robertson RM, Medina E, Shah N, Furlan R, Mosqueda-Garcia R. Neurally mediated syncope: pathophysiology and implications for treatment. Am J Med Sci. 1999 Feb;317(2):102-9. doi: 10.1097/00000441-199902000-00004. PMID 10037113
- [Background] Goldstein DS, Holmes C, Frank SM, Dendi R, Cannon RO 3rd, Sharabi Y, Esler MD, Eisenhofer G. Cardiac sympathetic dysautonomia in chronic orthostatic intolerance syndromes. Circulation. 2002 Oct 29;106(18):2358-65. doi: 10.1161/01.cir.0000036015.54619.b6. PMID 12403667
- [Background] Jacobs MC, Goldstein DS, Willemsen JJ, Smits P, Thien T, Dionne RA, Lenders JW. Neurohumoral antecedents of vasodepressor reactions. Eur J Clin Invest. 1995 Oct;25(10):754-61. doi: 10.1111/j.1365-2362.1995.tb01954.x. PMID 8557062